CLINICAL TRIAL: NCT01682603
Title: Effect of Botulinum Toxin A on Detrusor Overactivity and Renal Function in Chronic Spinal Cord Injured Patients - Clinical Effects and Investigating Mechanism of Action
Brief Title: Effect of Botulinum Toxin A on Detrusor Overactivity and Renal Function in Chronic Spinal Cord Injured Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Director of Urology, Buddhist Tzu Chi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCGHUROL005
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2014-06

CONDITIONS: Spinal Cord Injuries
Keywords: Nerve growth factor; P2X3 receptor; Transient Receptor Potential Vanilloid 1 (TRPV-1) receptor; Bladder function; Glomerular filtration rate; Detrusor overactivity; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Hereditary Sensory and Autonomic Neuropathies; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum toxin A (Experimental): BoNT-A (BOTOX 300U)
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — BoNT-A (BOTOX 300U)
  Other Names: BoNT-A (BOTOX 300U)

SUMMARY:
To investigate the clinical effect of detrusor botulinum toxin A (BoNT-A) injection on neurogenic detrusor overactivity (NDO) and renal function and to compare the difference of expressions of sensory receptors and nerve growth factor (NGF) in the bladder wall of patients respond and not respond to BoNT-A injections in chronic spinal cord injured (SCI) patients.

DETAILED DESCRIPTION:
Study Procedure

A total of 30 patients with chronic suprasacral cord SCI will be enrolled in this study. All patients are more than 18 years old and have chronic suprasacral cord injury for more than 1 year. They have previously underwent an urodynamic study and have been proven having detrusor sphincter dyssynergia (DSD). The patients currently void by reflex, abdominal stimulation or clean intermittent catheterization (CIC), are free of indwelling catheter or cystostomy, and free of urinary tract infection (UTI) on their enrollment. During the screening period, a total glomerular filtration rate (GFR) should be less than 80 mL/min as measured by 99mTc-labelled diethylenetriamine pentaacetic acid (99mTc-DTPA) clearance renal scanning. Patients should also have adequate hand function or have a care-giver available for CIC. Other exclusion criteria include patients with detrusor underactivity and large bladder compliance, patients proven to have intrinsic sphincteric deficiency and patients who have hypersensitivity to botulinum toxin A (BTX-A) or constituent ingredients of BTX-A.

BTX-A injection will be performed in the operation room under light intravenous general anesthesia to prevent autonomic dysreflexia and hyperreflexia during cystoscopy. A total of 300U BTX-A (BOTOX, 100 U/vial, Allergan Co., Irvine, USA) dissolved into 30 mL normal saline will be injected into 30 sites of the bladder including lateral, posterior wall and dome. The injection sites are widely distributed to cover the whole bladder wall. A 14 Fr Foley catheter will be routinely inserted after BTX-A injection and patients will be discharged the next morning and followed up at out-patient clinic. All patients will be instructed to keep on CIC or abdominal stimulation as they previously performed. BTX-A injections will be repeated 6 months after the first treatment, then follow up to 24 months. Before each BTX-A injection a videourodynamic study and GFR test will be performed. Patients were also requested to report the severity of urinary incontinence by the mean daily incontinence episodes within three days, Urogenital Distress Inventory (UDI-6 Short Form), Incontinence Impact Questionnaire (IIQ-7), self assessed QoL index and the global satisfaction rate (graded as 0 to 3, indicating none, mild, moderate and very satisfied) to this treatment. The adverse events such as urinary tract infection, hematuria, difficult urination are also recorded.

This study should be approved by the Institutional Review Board and Ethics Committee of the hospital. Informed consent will be obtained before the screening and all patients are instructed about the possible complications related with BTX-A injection such as urinary retention, transient hematuria and subsequent urinary tract infection.

Patients will be classified as responders and non-responders according to their clinical presentation and urodynamic study results. Responders are considered if they become dry or reduction of incontinence episodes by 50% and have a decrease of detrusor pressure reduction by 50% of the baseline value, otherwise, they are considered as non-responders. The end-point is set at 6 months after the BTX-A injection.

There were two primary end-points: (1) the net change of the IIQ-7 and UDI-6 from baseline to 24 months, and (2) the net change of the GFR from baseline to 24 months. Secondary end-point efficacy measured the net change of the cystometric bladder capacity, bladder compliance, detrusor pressure during reflex voiding, end-filling pressure or detrusor leak-point pressure and postvoid residual volume from baseline to 24 months.

Three bladder biopsies using a small cystoscopic biopsy forceps will be performed in all patients. The biopsy will be performed at baseline and each time-point just prior to intravesical BTX-A injection. The bladder biopsy specimens will be sent to pathological department for H-E staining to exclude the possibility of carcinoma in situ, and also will be embedded in O.C.T. medium and stored at -80℃ refrigerator or liquid nitrogen tank for investigations. The bladder biopsies will be prepared for measurement of NGF messenger RNA (mRNA) and immunohistochemistry investigation of the expression of Transient Receptor Potential Vanilloid 1 (TRPV-1), purinergic receptor P2X, ligand-gated ion channel, 3 (P2X3) receptors at baseline and 6 months after each BTX-A injection, and the difference of these sensory protein expressions between responders and .non-responders to BTX-A injection.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age of 19 years old or above
* Patients with chronic suprasacral cord SCI will be enrolled.
* Patients will be proven having NDO by videourodynamic study during the screening period.
* They also receive 99mTc-DTPA renal scanning for GFR at baseline.
* Patients with NDO induced urinary incontinence who have adequate hand function or have a care-giver available for CIC, and the baseline total GFR of less than 80 mL/min are main inclusion criteria

Exclusion Criteria:

* Patients with detrusor underactivity and large bladder compliance, patients proven to have intrinsic sphincteric deficiency
* Patients who have hypersensitivity to BTX-A or constituent ingredients of BTX-A.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

REFERENCES:
- [Background] Weld KJ, Graney MJ, Dmochowski RR. Clinical significance of detrusor sphincter dyssynergia type in patients with post-traumatic spinal cord injury. Urology. 2000 Oct 1;56(4):565-8. doi: 10.1016/s0090-4295(00)00761-5. PMID 11018603
- [Background] Ahmed HU, Shergill IS, Arya M, Shah PJ. Management of detrusor-external sphincter dyssynergia. Nat Clin Pract Urol. 2006 Jul;3(7):368-80. doi: 10.1038/ncpuro0521. PMID 16835625
- [Background] Weld KJ, Dmochowski RR. Association of level of injury and bladder behavior in patients with post-traumatic spinal cord injury. Urology. 2000 Apr;55(4):490-4. doi: 10.1016/s0090-4295(99)00553-1. PMID 10736489
- [Background] Linsenmeyer TA, Bagaria SP, Gendron B. The impact of urodynamic parameters on the upper tracts of spinal cord injured men who void reflexly. J Spinal Cord Med. 1998 Jan;21(1):15-20. doi: 10.1080/10790268.1998.11719505. PMID 9541882
- [Background] Ethans KD, Nance PW, Bard RJ, Casey AR, Schryvers OI. Efficacy and safety of tolterodine in people with neurogenic detrusor overactivity. J Spinal Cord Med. 2004;27(3):214-8. doi: 10.1080/10790268.2004.11753751. PMID 15478523
- [Background] Schurch B, Stohrer M, Kramer G, Schmid DM, Gaul G, Hauri D. Botulinum-A toxin for treating detrusor hyperreflexia in spinal cord injured patients: a new alternative to anticholinergic drugs? Preliminary results. J Urol. 2000 Sep;164(3 Pt 1):692-7. doi: 10.1097/00005392-200009010-00018. PMID 10953127
- [Background] Schulte-Baukloh H, Schobert J, Stolze T, Sturzebecher B, Weiss C, Knispel HH. Efficacy of botulinum-A toxin bladder injections for the treatment of neurogenic detrusor overactivity in multiple sclerosis patients: an objective and subjective analysis. Neurourol Urodyn. 2006;25(2):110-5. doi: 10.1002/nau.20153. PMID 16470519
- [Background] Schurch B, Hauri D, Rodic B, Curt A, Meyer M, Rossier AB. Botulinum-A toxin as a treatment of detrusor-sphincter dyssynergia: a prospective study in 24 spinal cord injury patients. J Urol. 1996 Mar;155(3):1023-9. doi: 10.1016/s0022-5347(01)66376-6. PMID 8583552
- [Background] Kuo HC. Botulinum A toxin urethral injection for the treatment of lower urinary tract dysfunction. J Urol. 2003 Nov;170(5):1908-12. doi: 10.1097/01.ju.0000091281.50081.f0. PMID 14532805
- [Background] Reitz A, Stohrer M, Kramer G, Del Popolo G, Chartier-Kastler E, Pannek J, Burgdorfer H, Gocking K, Madersbacher H, Schumacher S, Richter R, von Tobel J, Schurch B. European experience of 200 cases treated with botulinum-A toxin injections into the detrusor muscle for urinary incontinence due to neurogenic detrusor overactivity. Eur Urol. 2004 Apr;45(4):510-5. doi: 10.1016/j.eururo.2003.12.004. PMID 15041117
- [Background] Kuo HC. Therapeutic effects of suburothelial injection of botulinum a toxin for neurogenic detrusor overactivity due to chronic cerebrovascular accident and spinal cord lesions. Urology. 2006 Feb;67(2):232-6. doi: 10.1016/j.urology.2005.08.016. Epub 2006 Jan 25. PMID 16442605
- [Background] Schulte-Baukloh H, Weiss C, Stolze T, Herholz J, Sturzebecher B, Miller K, Knispel HH. Botulinum-A toxin detrusor and sphincter injection in treatment of overactive bladder syndrome: objective outcome and patient satisfaction. Eur Urol. 2005 Dec;48(6):984-90; discussion 990. doi: 10.1016/j.eururo.2005.06.021. Epub 2005 Jul 18. PMID 16126328
- [Background] Schurch B, de Seze M, Denys P, Chartier-Kastler E, Haab F, Everaert K, Plante P, Perrouin-Verbe B, Kumar C, Fraczek S, Brin MF; Botox Detrusor Hyperreflexia Study Team. Botulinum toxin type a is a safe and effective treatment for neurogenic urinary incontinence: results of a single treatment, randomized, placebo controlled 6-month study. J Urol. 2005 Jul;174(1):196-200. doi: 10.1097/01.ju.0000162035.73977.1c. PMID 15947626
- [Background] Grosse J, Kramer G, Stohrer M. Success of repeat detrusor injections of botulinum a toxin in patients with severe neurogenic detrusor overactivity and incontinence. Eur Urol. 2005 May;47(5):653-9. doi: 10.1016/j.eururo.2004.11.009. Epub 2005 Jan 15. PMID 15826758
- [Background] Yiangou Y, Facer P, Ford A, Brady C, Wiseman O, Fowler CJ, Anand P. Capsaicin receptor VR1 and ATP-gated ion channel P2X3 in human urinary bladder. BJU Int. 2001 Jun;87(9):774-9. doi: 10.1046/j.1464-410x.2001.02190.x. PMID 11412212
- [Background] Wiseman OJ, Fowler CJ, Landon DN. The role of the human bladder lamina propria myofibroblast. BJU Int. 2003 Jan;91(1):89-93. doi: 10.1046/j.1464-410x.2003.03802.x. PMID 12614258
- [Background] Cockayne DA, Hamilton SG, Zhu QM, Dunn PM, Zhong Y, Novakovic S, Malmberg AB, Cain G, Berson A, Kassotakis L, Hedley L, Lachnit WG, Burnstock G, McMahon SB, Ford AP. Urinary bladder hyporeflexia and reduced pain-related behaviour in P2X3-deficient mice. Nature. 2000 Oct 26;407(6807):1011-5. doi: 10.1038/35039519. PMID 11069181
- [Background] Avelino A, Cruz C, Nagy I, Cruz F. Vanilloid receptor 1 expression in the rat urinary tract. Neuroscience. 2002;109(4):787-98. doi: 10.1016/s0306-4522(01)00496-1. PMID 11927161
- [Background] Namasivayam S, Eardley I, Morrison JF. Purinergic sensory neurotransmission in the urinary bladder: an in vitro study in the rat. BJU Int. 1999 Nov;84(7):854-60. doi: 10.1046/j.1464-410x.1999.00310.x. PMID 10532986
- [Background] Morrison J, Wen J, Kibble A. Activation of pelvic afferent nerves from the rat bladder during filling. Scand J Urol Nephrol Suppl. 1999;201:73-5. PMID 10573780
- [Background] Gabella G. The structural relations between nerve fibres and muscle cells in the urinary bladder of the rat. J Neurocytol. 1995 Mar;24(3):159-87. doi: 10.1007/BF01181533. PMID 7798112
- [Background] Aoki KR. Evidence for antinociceptive activity of botulinum toxin type A in pain management. Headache. 2003 Jul-Aug;43 Suppl 1:S9-15. doi: 10.1046/j.1526-4610.43.7s.3.x. PMID 12887389
- [Background] Durham PL, Cady R, Cady R. Regulation of calcitonin gene-related peptide secretion from trigeminal nerve cells by botulinum toxin type A: implications for migraine therapy. Headache. 2004 Jan;44(1):35-42; discussion 42-3. doi: 10.1111/j.1526-4610.2004.04007.x. PMID 14979881
- [Background] Cruz F, Guimaraes M, Silva C, Reis M. Suppression of bladder hyperreflexia by intravesical resiniferatoxin. Lancet. 1997 Aug 30;350(9078):640-1. doi: 10.1016/S0140-6736(05)63330-2. No abstract available. PMID 9288055
- [Background] Apostolidis A, Popat R, Yiangou Y, Cockayne D, Ford AP, Davis JB, Dasgupta P, Fowler CJ, Anand P. Decreased sensory receptors P2X3 and TRPV1 in suburothelial nerve fibers following intradetrusor injections of botulinum toxin for human detrusor overactivity. J Urol. 2005 Sep;174(3):977-82; discussion 982-3. doi: 10.1097/01.ju.0000169481.42259.54. PMID 16094018
- [Background] Fowler CJ, Beck RO, Gerrard S, Betts CD, Fowler CG. Intravesical capsaicin for treatment of detrusor hyperreflexia. J Neurol Neurosurg Psychiatry. 1994 Feb;57(2):169-73. doi: 10.1136/jnnp.57.2.169. PMID 8126498
- [Background] Silva C, Rio ME, Cruz F. Desensitization of bladder sensory fibers by intravesical resiniferatoxin, a capsaicin analog: long-term results for the treatment of detrusor hyperreflexia. Eur Urol. 2000 Oct;38(4):444-52. doi: 10.1159/000020322. PMID 11025384
- [Background] Giannantoni A, Di Stasi SM, Stephen RL, Bini V, Costantini E, Porena M. Intravesical resiniferatoxin versus botulinum-A toxin injections for neurogenic detrusor overactivity: a prospective randomized study. J Urol. 2004 Jul;172(1):240-3. doi: 10.1097/01.ju.0000132152.53532.5d. PMID 15201783
- [Background] Giannantoni A, Di Stasi SM, Nardicchi V, Zucchi A, Macchioni L, Bini V, Goracci G, Porena M. Botulinum-A toxin injections into the detrusor muscle decrease nerve growth factor bladder tissue levels in patients with neurogenic detrusor overactivity. J Urol. 2006 Jun;175(6):2341-4. doi: 10.1016/S0022-5347(06)00258-8. PMID 16697870
- [Background] Patel AK, Patterson JM, Chapple CR. Botulinum toxin injections for neurogenic and idiopathic detrusor overactivity: A critical analysis of results. Eur Urol. 2006 Oct;50(4):684-709; discussion 709-10. doi: 10.1016/j.eururo.2006.07.022. Epub 2006 Aug 4. PMID 16934391
- [Background] Kuo HC. Urodynamic evidence of effectiveness of botulinum A toxin injection in treatment of detrusor overactivity refractory to anticholinergic agents. Urology. 2004 May;63(5):868-72. doi: 10.1016/j.urology.2003.12.007. PMID 15134967
- [Background] Steers WD. Pathophysiology of overactive bladder and urge urinary incontinence. Rev Urol. 2002;4 Suppl 4(Suppl 4):S7-S18. PMID 16986023
- [Background] Chartier-Kastler E, Comperat E, Ruffion A. [Disorders of bladder compliance and neurogenic bladder]. Prog Urol. 2007 May;17(3):442-7. doi: 10.1016/s1166-7087(07)92345-3. French. PMID 17622074
- [Background] Sekar P, Wallace DD, Waites KB, DeVivo MJ, Lloyd LK, Stover SL, Dubovsky EV. Comparison of long-term renal function after spinal cord injury using different urinary management methods. Arch Phys Med Rehabil. 1997 Sep;78(9):992-7. doi: 10.1016/s0003-9993(97)90063-0. PMID 9305274
- [Background] Gerridzen RG, Thijssen AM, Dehoux E. Risk factors for upper tract deterioration in chronic spinal cord injury patients. J Urol. 1992 Feb;147(2):416-8. doi: 10.1016/s0022-5347(17)37254-3. PMID 1732606
- [Background] Weld KJ, Graney MJ, Dmochowski RR. Differences in bladder compliance with time and associations of bladder management with compliance in spinal cord injured patients. J Urol. 2000 Apr;163(4):1228-33. PMID 10737503
- [Background] Giannantoni A, Scivoletto G, Di Stasi SM, Silecchia A, Finazzi-Agro E, Micali I, Castellano V. Clean intermittent catheterization and prevention of renal disease in spinal cord injury patients. Spinal Cord. 1998 Jan;36(1):29-32. doi: 10.1038/sj.sc.3100509. PMID 9471135
- [Background] Pannek J, Sommerfeld HJ, Botel U, Senge T. Combined intravesical and oral oxybutynin chloride in adult patients with spinal cord injury. Urology. 2000 Mar;55(3):358-62. doi: 10.1016/s0090-4295(99)00540-3. PMID 10699610
- [Background] Nosseir M, Hinkel A, Pannek J. Clinical usefulness of urodynamic assessment for maintenance of bladder function in patients with spinal cord injury. Neurourol Urodyn. 2007;26(2):228-33. doi: 10.1002/nau.20319. PMID 16998859
- [Background] Razdan S, Leboeuf L, Meinbach DS, Weinstein D, Gousse AE. Current practice patterns in the urologic surveillance and management of patients with spinal cord injury. Urology. 2003 May;61(5):893-6. doi: 10.1016/s0090-4295(02)02518-9. PMID 12735998
- [Background] MacDiarmid SA, McIntyre WJ, Anthony A, Bailey RR, Turner JG, Arnold EP. Monitoring of renal function in patients with spinal cord injury. BJU Int. 2000 Jun;85(9):1014-8. doi: 10.1046/j.1464-410x.2000.00680.x. PMID 10848686
- [Background] Samson G, Cardenas DD. Neurogenic bladder in spinal cord injury. Phys Med Rehabil Clin N Am. 2007 May;18(2):255-74, vi. doi: 10.1016/j.pmr.2007.03.005. PMID 17543772
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Chan CL, Facer P, Davis JB, Smith GD, Egerton J, Bountra C, Williams NS, Anand P. Sensory fibres expressing capsaicin receptor TRPV1 in patients with rectal hypersensitivity and faecal urgency. Lancet. 2003 Feb 1;361(9355):385-91. doi: 10.1016/s0140-6736(03)12392-6. PMID 12573376
- [Background] Shu SY, Ju G, Fan LZ. The glucose oxidase-DAB-nickel method in peroxidase histochemistry of the nervous system. Neurosci Lett. 1988 Feb 29;85(2):169-71. doi: 10.1016/0304-3940(88)90346-1. PMID 3374833
- [Background] Schrader AJ, Lauber J, Lechner O, Heidenreich A, Hofmann R, Buer J. Application of real-time reverse transcriptase-polymerase chain reaction in urological oncology. J Urol. 2003 May;169(5):1858-64. doi: 10.1097/01.ju.0000047363.03411.6b. PMID 12686862
- [Background] Yono M, Takahashi W, Pouresmail M, Johnson DR, Foster HE Jr, Weiss RM, Latifpour J. Quantification of endothelins, their receptors, and endothelin-converting enzyme mRNAs in rat genitourinary tract using real-time RT-PCR. J Pharmacol Toxicol Methods. 2002 Sep-Oct;48(2):87-95. doi: 10.1016/s1056-8719(03)00022-4. PMID 14565565
- [Background] Cruz F, Avelino A, Cruz C, et al. Sensory fibers immunoreactive to the vanilloid receptor protein: Distribution in the urinary bladder. Neurourol Urodynam 19:456, 2000.
- [Background] Cui M, Aoki KR. Botulinum toxin type A(BTX-A) reduces inflammatory pain in the rat formalin model. Cephalalgia 20:414, 2000.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The chronic SCI patients with urinary incontinence in Hualien Tzu Chi General Hospital were consecutively recruited into this study.
Pre-assignment Details: Patients were excluded if they had an active urinary tract infection, urinary tract cancer, history of lower urinary tract surgery or chronic systemic diseases. If patients fulfilled the inclusion criteria, they were enrolled in this study.
Groups:
- Botulinum Toxin A: Botulinum toxin A (BoNT-A) (BOTOX 300U)
Period: Overall Study
Arm/Group | Botulinum Toxin A
Started | 37
Completed | 34
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 41.5 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Region of Enrollment [Number; unit: participants]
  Taiwan | 34
Injury Level [Number; unit: participants]
  Cervical | 13
  Thoracic | 21
ASIA Classification [Number; unit: participants] — ASIA Impairment Scale A: Complete. No sensory or motor function is preserved in the sacral segments S4-S5. B: Incomplete. Sensory but not motor function is preserved below the neurological level and includes the sacral segments S4-S5. C: Incomplete. Motor function is preserved below the neurological level, and more then half of key muscles below the neurological level have a muscle grade less then 3 (Grades 0-2). D: Incomplete. Motor function is preserved below the neurological level, and at least half of key muscles below the neurological level have a muscle grade greater than or equal to 3.
  participants
    A | 27
    B | 3
    C | 2
    D | 2
Autonomic dysreflexia [Number; unit: participants]
  Autonomic dysreflexia | 11
  Non-Autonomic dysreflexia | 23

OUTCOME MEASURES:

1. Primary Outcome: Net Change of the Urinary Distress Inventory (UDI-6)
Description: Efficacy:
  Net change of the UrinaryDdistress Inventory (UDI-6) from baseline and 12 months.
  The UDI-6 is a 6-item short forms on a 4-point scale ranging from 0 "Not at all" to 3 "Greatly".
  The total UDI-6 score can therefore range from 0 to 18 (asymptomatic to very symptomatic).
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
units on a scale
  Baseline | 10.4 (4.13)
  12 months | 7.43 (2.24)

2. Secondary Outcome: Net Change of the Cystometric Bladder Capacity (CBC)
Description: Efficacy:
  Net change of the cystometric bladder capacity (CBC) from baseline and 12 months
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
mL
  Baseline | 305.9 (167.7)
  12 months | 437.6 (114.3)

3. Secondary Outcome: Net Change of the Bladder Compliance
Description: Bladder compliance is the result of a mathematical calculation of the volume required for a unit rise of pressure measured during a cystometric filling.
  Bladder compliance is calculated by dividing the volume change by the change in bladder pressure (mL/cmH2O).
  Efficacy:
  Net change of the bladder compliance from baseline and 12 months
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
mL/cmH2O
  Baseline | 30.6 (29.1)
  12 months | 29.0 (19.6)

4. Secondary Outcome: Net Change of the Maximum Flow Rate (Qmax)
Description: Efficacy:
  Net change of the maximum flow rate (Qmax) from baseline and 12 months
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
mL/s
  Baseline | 4.56 (4.75)
  12 months | 3.54 (8.85)

5. Secondary Outcome: Net Change of the Void Volume
Description: Efficacy:
  Net change of the void volume from baseline and 12 months
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
mL
  Baseline | 79.6 (95.1)
  12 months | 59.2 (125.1)

6. Secondary Outcome: Net Change of the Detrusor Pressure (Pdet)
Description: Efficacy:
  Net change of the detrusor pressure (Pdet) from baseline and 12 months
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
cmH2O
  Baseline | 36.1 (22.2)
  12 months | 12.9 (16.9)

7. Secondary Outcome: Net Change of the Postvoid Residual Volume (PVR)
Description: Efficacy:
  Net change of the postvoid residual volume (PVR) from baseline and 12 months
  Results:
  Botulinum toxin A injection have increased postvoid residual urine volume in patients treated for bladder dysfunction.
  Treat only patients who are willing and able to initiate catheterization post-treatment, if required, for urinary retention.
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
mL
  Baseline | 226.3 (138.2)
  12 months | 378.5 (142.1)

8. Primary Outcome: Net Change of the Incontinence Impact Questionnaire (IIQ-7)
Description: Efficacy:
  Net change of the Incontinence Impact Questionnaire (IIQ-7) from baseline and 12 months.
  The IIQ-7 is a 7-item short forms on a 4-point scale ranging from 0 "Not at all" to 3 "Greatly".
  Total IIQ-7 score ranges = 0 to 21 The total IIQ-7 score can therefore range from 0 to 21 (asymptomatic to very symptomatic).
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
units on a scale
  Baseline | 11.9 (5.22)
  12 months | 5.57 (4.97)

9. Primary Outcome: Net Change of the Quality of Life Index (QoL-I)
Description: Efficacy:
  Net change of the quality of life index (QoL-I) from baseline and 12 months. The QoL-I on a 7-point scale ranging from 0 "Delighted" to 6 "Terrible". The QoL-I ranges 0 to 6
  Safety:
  Systemic adverse events
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A
Number analyzed (Participants) | 34
units on a scale
  Baseline | 4.00 (1.24)
  12 months | 2.21 (1.48)

10. Other Pre Specified Outcome: Autonomic Dysreflexia
Time Frame: Baseline and 12 months
Measure: Number; unit: participants
Groups:
- Pre-Autonomic Dysreflexia: Baseline Autonomic dysreflexia
- Pre-Non Autonomic Dysreflexia: Baseline Non autonomic dysreflexia
Arm/Group | Pre-Autonomic Dysreflexia | Pre-Non Autonomic Dysreflexia
Number analyzed (Participants) | 11 | 23
participants
  Post-Autonomic dysreflexia | 5 | 1
  Post-Non Autonomic dysreflexia | 6 | 22

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Botulinum Toxin A
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 22/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin A (N=34)
De nove autonomic dysreflexia (Nervous system disorders) | 6
Difficult urination (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Urinary tract infection (Renal and urinary disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes